CLINICAL TRIAL: NCT05503914
Title: Sichuan Cancer Hospital and Institute, Sichuan Cancer Center, School of Medicine, University of Electronic Science and Technology of China
Brief Title: Low-dose Radiotherapy and Neoadjuvant Chemotherapy Sequential Concurrent Chemoradiotherapy for Locally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Mei Feng, Vice President, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahead-NC-202208
Record Dates: First submitted 2022-08-12; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose radiotherapy group (Experimental): Neoadjuvant chemotherapy combined with low-dose radiotherapy sequential concurrent chemoradiotherapy
  Interventions: Radiation: low-dose radiotherapy
- control group (No Intervention): Neoadjuvant chemotherapy sequential concurrent chemoradiotherapy

INTERVENTIONS:
Radiation: low-dose radiotherapy — On the first and second days of induction chemotherapy, local tumor were irradiated with 0.5Gy bid for 4 times.
  Arms: low-dose radiotherapy group

SUMMARY:
Nasopharyngeal carcinoma#NPC#is common malignant tumor in China. The incidence of NPC in most parts of the world and the country is less than 1/10 million, but the incidence rate in China's Guangdong, Guangxi, Fujian and other southern provinces is as high as 33/10 million. Generally, there are more men than women, with a ratio of 2 ~ 3:1. In high incidence area, nasopharyngeal carcinoma has great harm to middle-aged and young people, and incidence rate and mortality rate increase significantly after 30 years old. 50~60 years old is the highest peak. More than 70% of patients were in advanced stage at the first diagnosis. At present, the main treatment for locally advanced nasopharyngeal carcinoma is platinum based neoadjuvant chemotherapy combined with concurrent chemoradiotherapy. However, recurrence and distant metastasis after standard treatment are the main causes of failure. About 40% of patients with locally advanced nasopharyngeal carcinoma have recurrence and distant metastasis after receiving standard treatment. Therefore, the investigators intend to further explore the improvement of local control and survival rate of locally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma NPC is common malignant tumor in China. The incidence of NPC in most parts of the world and the country is less than 1/10 million, but the incidence rate in China's Guangdong, Guangxi, Fujian and other southern provinces is as high as 33/10 million. According to the statistics of the international cancer research center, there were about 129000 new cases of nasopharyngeal carcinoma in 2018.The pathogenesis of NPC is caused by many factors: heredity, environment and virus infection. Among them, EB virus is closely related to the pathogenesis of NPC. Generally, there are more men than women, with a ratio of 2 ~ 3:1. In high incidence area, nasopharyngeal carcinoma has great harm to middle-aged and young people, and incidence rate and mortality rate increase significantly after 30 years old. 50~60 years old is the highest peak. More than 70% of patients were in advanced stage at the first diagnosis. At present, the main treatment for locally advanced nasopharyngeal carcinoma is platinum based neoadjuvant chemotherapy combined with concurrent chemoradiotherapy. Radiotherapy is the main treatment of nasopharyngeal carcinoma. With the application of intensity modulated radiotherapy, the 5- year local control and regional recurrence free survival rate of nasopharyngeal carcinoma have been increased to more than 83%. However, recurrence and distant metastasis after standard treatment are the main causes of failure. About 40% of patients with locally advanced nasopharyngeal carcinoma have recurrence and distant metastasis after receiving standard treatment.A large number of clinical studies and meta-analysis show that induction chemotherapy combined with concurrent chemoradiotherapy can significantly improve the progression free survival rate and overall survival rate compared with concurrent chemoradiotherapy alone. Induction chemotherapy can reduce the risk of systemic recurrence and metastasis by controlling the occurrence of tumor. Based on the above research, neoadjuvant chemotherapy for locally advanced nasopharyngeal carcinoma has been written into the national comprehensive cancer network(NCCN) of the United States and the Chinese Clinical Oncology(CSCO) guidelines.In recent years, a large number of studies are exploring various radiotherapy strategies, such as changing the mode of radiotherapy segmentation and hypersensitivity (HRS), in order to further improve local control and survival.Therefore, the investigators plan to carry out a randomized, controlled phase II prospective clinical study of neoadjuvant chemotherapy combined with low-dose radiotherapy and sequential concurrent radiotherapy and chemotherapy in the treatment of locally advanced nasopharyngeal carcinoma.

Joiner recognized the potential of low-dose fractionated radiotherapy as early as 20 years ago. Namely: high radiosensitivity (HRS), which means that the initial dose can produce radiosensitivity from 0 to 80 cGy. Low-dose fractionated radiation therapy (LDFRT) is a unique radiobiological phenomenon. This phenomenon reports that the effect of induced chemotherapy can be increased by reducing MDR-1 and overcoming the antiapoptotic effect of Bcl-2, resulting in the death of nuclear factors kappa-b29 and p53.This radiation is different from conventional fractionated or large fractionated radiotherapy. Conventional segmentation or high-dose segmentation will not only kill tumor cells, but also make tumor cells resistant to radiation. Studies have shown that low-dose radiotherapy (LDFRT) in the range of 50 - 80 cGy can be used as a chemical sensitizer to enhance the effect of chemotherapy, increase tumor response and improve local control. At present, clinical studies have reported that in locally advanced Squamous cell carcinoma of head and neck#SCCHN#, the clinical experiment of induction chemotherapy (paclitaxel + carboplatin) combined with LDFRT has achieved preliminary success, and showed that the optimal dose is 50-80cGy 4 times / day. Importantly, it did not increase the toxic and side effects of induction chemotherapy. Subsequently, the results of a long-term SCCHN trial reported that the primary endpoint complete response rate (CR), secondary endpoint overall survival (OS), progression free survival (PFS) and toxicity of LDFRT combined with induction chemotherapy had clinical significance. At present, the role of LDFRT in locally advanced nasopharyngeal carcinoma is still unclear. Whether it can improve the efficacy of neoadjuvant chemotherapy is worth exploring.

In conclusion, neoadjuvant chemotherapy combined with LDFRT provides a new idea for tumor treatment. Low dose fractionated radiotherapy is used to enhance the objective remission rate of induction chemotherapy, make high-risk tumor lesions become the target area, and up regulate the apoptotic proteins bax and bcl-x in the microenvironment to achieve the greatest benefit. Therefore, it is of great clinical value to explore the application of neoadjuvant chemotherapy combined with low-dose radiotherapy (LDFRT) sequential concurrent chemoradiotherapy in locally advanced nasopharyngeal carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate and sign the informed consent form of the study in writing 2. Age 18-70 years old, regardless of gender 3. Pathological biopsy confirmed nasopharyngeal squamous cell carcinoma 4. Initial treatment 5. There are lesions that can be measured according to RECIST standard 6. KPS score ≥ 80 7. Estimated survival ≥ 6 months 8. The urine pregnancy test was negative (female), and contraceptive measures were taken from the test period to 3 months after the end of the test 9. Sufficient hematopoietic function: WBC ≥ 4 × 109/L#Hb≥100g/ L#PLT≥100 × 109/L 10. Liver function: ALAT / ASAT < 1.5 times of ULN, bilirubin < 1.5 × ULN 11. Renal function: serum creatinine < 1.5 × ULN 12. No distant metastasis 13.T3-T4 (AJCC / UICC 8th Edition) nasopharyngeal carcinoma 14. According to the judgment of the researcher, the patient is considered to be able to comply with the protocol.

Exclusion Criteria:

1. Those who have received epidermal growth factor targeted therapy
2. The primary focus has received immunotherapy
3. Other malignant tumors (except non melanoma skin cancer or cervical carcinoma in situ)
4. Subjects who have received other drug trials in recent 1 month
5. Have a serious history of allergy or special constitution
6. A history of severe lung or heart disease or serious complications, such as uncontrollable hypertension and heart failure.
7. Drug or alcohol addicts
8. Having personality or mental illness, no civil capacity or limited civil capacity
9. Active systemic infection
10. At the same time, they received chronic systemic immunotherapy or hormone therapy other than this study. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
The objective remission rate | assessed up to 1 month
  The main indicator is objective remission rate (ORR=CR+PR)

SECONDARY OUTCOMES:
Adverse events and reactions | assessed up to 1 month
  evaluated according to NCI CTCAE version 3.0 Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: feng mei, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Low-dose Radiotherapy and Neoadjuvant Chemotherapy Sequential Concurrent Chemoradiotherapy for Locally Advanced Nasopharyngeal Carcinoma, Sichuan, Sichuan, China